CLINICAL TRIAL: NCT05614778
Title: A Multicenter, Noninterventional, Prospective Study to Investigate the Efficacy and Safety After Administration of Daewoong Zoledronic Acid for the Purpose of Treatment or Prevention of Osteoporosis in Real-world Observational Study
Brief Title: Study to Investigate the Efficacy and Safety After Administration of Daewoong Zoledronic Acid for the Purpose of Treatment or Prevention of Osteoporosis
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWZA_OS01
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment group: Zoledronic Acid inj. 5mg/100mL
  Interventions: Other: Zoledronic Acid injection, 5mg/100mL

INTERVENTIONS:
Other: Zoledronic Acid injection, 5mg/100mL — Zoledronic Acid injection, 5mg/100mL

SUMMARY:
This study is a non-interventional observational study. On the baseline (Visit 1), we collect demographic data from all participating subjects according to their daily medical conditions, prescribe drugs and collect validity and safety data according to the research plan in Visit 1 and Visit 2. In addition, we collect data by application on subject's self-awareness symptoms and subject's questionnaire for medical outcome short form health survey (SF-36) every day from the baseline for 4 days.

DETAILED DESCRIPTION:
The investigator will enroll subjects according to Inclusion/Exclusion criteria after obtaining Informed Consent Form from each subject. Enrolled subjects will administer Zoledronic Acid 5mg/100mL once on baseline (Visit 1). The demographic data, prescription data, and medical history, etc will be collected based on the approved protocol. Additionally using application, subject's self-awareness symptoms and subject's questionnaire for medical outcome short form health survey (SF-36) every day from the baseline for 4 days will be collected.

Investigator will also collect any occurrence of fracture through electronic medical record until 48 weeks (Visit 2) from baseline visit.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults 19 years of age or older at the time of screening visit
2. A person who is scheduled to administer the research drug according to the medical judgment of the researcher based on the permission
3. A person who can understand the information provided to the person and can voluntarily sign a written consent form

Exclusion Criteria:

1. Those subject to contraindications to administration according to the drug approval requirements for research

   * Patients with hypersensitivity to the components of this drug or other bisphosphonate drugs Hypocalcemia
   * Patients with severe renal impairment whose creatinine clearance rate is less than 35 mL/min (patients must measure serum creatinine and creatinine clearance before receiving the study drug).
   * Patients receiving Zometa for cancer as an indication
   * Pregnant women, women who may be pregnant, and lactating women
2. Patients participating in other clinical trials (However, registration is possible if you have not received investigational drugs or are participating in other non-interventional observational studies.)
3. In addition to the above, patients whom the researcher (physician in charge) determines are not suitable as subjects of this observational study.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Study population was calculated by using PASS16, Confidence intervals for one mean procedure.
Sampling Method: Probability Sample
Enrollment: 2881 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Lumbar spine bone mineral density (BMD) change rate | 48 weeks
  Lumbar spine bone mineral density (BMD) change rate at 48 weeks compared to baseline

SECONDARY OUTCOMES:
Changes in lumbar spine, femur, hip joint, and bone mineral density (BMD) | 48 weeks
  Changes in lumbar spine, femur, hip joint, and bone mineral density (BMD) at 48 weeks compared to baseline
New clinical fracture incidence | 48 weeks
  New clinical fracture incidence at 48 weeks (%)
Investigator satisfaction score | 48 weeks
  Investigator satisfaction score at 48 weeks
Safety evaluation | 48 weeks
  Safety evaluation related to Daewoong zoledronic acid administration

CONTACTS AND LOCATIONS:
Overall Officials: Yumie Lee, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided